CLINICAL TRIAL: NCT03020199
Title: A Randomized, Multicenter STudy to Evaluate the Effect of Secukinumab 300 mg s.c. Administered During 52 Weeks to Patients Suffering From New-onset Moderate to Severe Plaque Psoriasis as Early Intervention Compared to Standard Treatment With Narrow-band UVB (STEPIn Study)
Brief Title: Study of the Efficacy of Early Intervention With Secukinumab 300 mg s.c. Compared to Narrow-band UVB in Patients With New-onset Moderate to Severe Plaque Psoriasis
Acronym: STEPin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAIN457A2322; 2015-002423-26 (EudraCT Number)
Record Dates: First submitted 2016-09-23; First posted 2017-01-13 (Estimated); Results first posted 2024-10-01 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Plaque Psoriasis
Keywords: Psoriasis; interleukin (IL) 17A; IL-17A; secukinumab; AIN457; Narrow-band ultraviolet light B; nb-UVB; Psoriasis area and severity index; PASI
MeSH Terms: conditions — Psoriasis | interventions — secukinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Secukinumab 300 mg (Experimental): In the Main Study, 80 new-onset psoriasis patients in Arm A1 (68 in Arm A1a, 12 in Arm A1b) received 300 mg secukinumab injections weekly for the first month, then every 4 weeks until Week 48 (52-week treatment). Arm A1b patients also joined the Mechanistic Sub-study.
  In the Mechanistic Sub-study, 12 new-onset psoriasis patients (Arm A2) and 24 chronic plaque psoriasis patients (12 each in Arms C1 and C2) received similar secukinumab treatment. Arm A2 and C2 patients continued until Week 100 (104-week treatment), while Arm C1 ended at Week 48 (52-week treatment).
  Interventions: Biological: Secukinumab
- Narrow-band ultraviolet B (nb-UVB) (Active Comparator): In the Main Study, 80 new-onset psoriasis patients in Arm B1 (68 in Arm B1a and 12 in Arm B1b) received 1 or 2 cycles of nb UVB of 12 weeks each with a maximum break of 28 weeks between cycles (patients with PASI 90 at Week 40 did not receive a second treatment cycle) (treatment duration = 52 weeks).
  Patients from Arm B1b participated also in the Mechanistic Sub-study.
  Interventions: Radiation: nb-UVB

INTERVENTIONS:
Biological: Secukinumab — Secukinumab (AIN457) 300 mg was administered in an open-label fashion according to label as 2 s.c. injections of secukinumab 150 mg (1-mL liquid formulation in a pre-filled syringe). Each 300-mg dose was provided as 2 pre-filled syringes of 150-mg secukinumab in a single box. Each syringe was labeled as AIN457 150 mg/1 mL.
  Other Names: AIN457
  Arms: Secukinumab 300 mg
Radiation: nb-UVB — Narrow-band UVB applied in 1 or 2 cycles, each comprising a period of 12 weeks with 2 to 3 treatment sessions per week totaling 24 to 36 sessions per cycle. The application was performed according to the investigational site's protocol, taking into account the patient's skin type. A maximum dose of 3 J/cm2 on the body and 1 J/cm2 on the face was recommended
  Arms: Narrow-band ultraviolet B (nb-UVB)

SUMMARY:
The purpose of this study was to determine whether early intervention with subcutaneous (s.c.) secukinumab 300 mg in patients with new-onset moderate to severe plaque psoriasis may lead to prolonged symptom-free periods by preventing reactivation of old lesions or ultimately totally hindering the occurrence of new lesions, i.e., changing the natural course of the disease (Main Study).

DETAILED DESCRIPTION:
This was and open label, parallel group, multicenter, randomized study with 3 clinical periods: Screening period, Treatment period, and Follow-up period.

The design consisted of the Main Study and a Mechanistic Sub study:

1. The Main Study had 2-treatment-arm secukinumab and nb-UVB).
2. The Mechanistic Sub-study had 4 arms treated with secukinumab and one arm with nb-UVB arm. The outcome measures were all exploratory, i.e. no results presented. Not all participants of the Mechanistic Sub-study participated in the Main Study, these participants are only reported for the safety analyses, but not for the primary and secondary outcome measures.

ELIGIBILITY:
Key Inclusion Criteria:

* Able to understand and communicate with the investigator, willing and capable to comply with all study procedures, and provide written signed and dated informed consent (personally or by a witness) before any assessment is performed.
* Aged 18 to 50 years inclusive.
* New-onset plaque psoriasis with appearance of the first psoriasis plaques within the last 12 months before randomization and naïve to any systemic treatment and phototherapy (Arm A1, Arm A2, and Arm B1). Episodes of mild psoriasis, which occurred at least 3 years before screening and resolved spontaneously within 6 months will be accepted.
* Chronic plaque psoriasis with appearance of the first psoriasis symptoms 5 years or longer and intolerance or inadequate response to phototherapy or any systemic treatment including biologicals, except for IL-17A inhibitors (Arm C1 and Arm C2).
* Moderate to severe plaque psoriasis defined at screening and baseline by PASI >= 10, and body surface area (BSA) >= 10%, and IGA mod 2011 >= 3.

Key Exclusion Criteria:

* Forms of psoriasis other than plaque-type (e.g., pustular, erythrodermic, guttate, light sensitive, and drug induced).
* Ongoing use of prohibited treatments.
* Previous treatment with phototherapy or any systemic treatment.
* Pregnant or nursing (lactating) women.
* Women of childbearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception during the Treatment period or longer if required by locally approved prescribing information (e.g., 20 weeks in the EU and countries where applicable for secukinumab).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 196 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2023-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (36):
- Argentina (2):
  - Novartis Investigative Site, Ciudad Autonoma de Bs As, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
- Bulgaria (3):
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
- Canada (2):
  - Novartis Investigative Site, Greater Sudbury, Ontario
  - Novartis Investigative Site, Markham, Ontario
- Novartis Investigative Site, Aarhus N, Denmark
- Estonia (2):
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- Finland (2):
  - Novartis Investigative Site, Tampere
  - Novartis Investigative Site, Turku
- Germany (3):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Frankfurt
- Hungary (2):
  - Novartis Investigative Site, Nyíregyháza
  - Novartis Investigative Site, Szolnok
- Poland (5):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lodz
- Spain (7):
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Alcorcón, Madrid
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Las Palmas de Gran Canaria
  - Novartis Investigative Site, Madrid
- Sweden (2):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Malmo
- Novartis Investigative Site, Lausanne, Switzerland
- United Kingdom (4):
  - Novartis Investigative Site, Bradford, West Yorkshire
  - Novartis Investigative Site, Leeds, West Yorkshire
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Salford

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled in 2 study sites in Argentina, 4 in Bulgaria, 2 in Canada, 4 in Germany, 1 in Denmark, 3 in Estonia, 2 in Finland, 2 in Hungary, 6 in Poland, 8 in Spain, 2 in Sweden, 1 in Switzerland, and 4 in the United Kingdom.
Groups:
- Secukinumab 300 mg: Eligible patients received 300 mg secukinumab by subcutaneous (s.c.) injection at baseline, Weeks 1, 2, 3, 4 and then every 4 weeks until Week 48 inclusive (treatment duration = 52 weeks) OR every 4 weeks until Week 100 inclusive (last dose administered at Week 100) (treatment duration = 104 weeks).
- Narrow-band Ultraviolet B (Nb-UVB): Eligible patients received 1 or 2 cycles of narrow-band ultraviolet B (nb-UVB) of 12 weeks each with a maximum break of 28 weeks between cycles (patients with PASI 90 at Week 40 will not receive a second treatment cycle) (treatment duration = 52 weeks).
Period: Treatment Period
Arm/Group | Secukinumab 300 mg | Narrow-band Ultraviolet B (Nb-UVB)
Started (All the subjects in the study were included in the Randomized Set and the Full Analysis Set (FAS).) | 116 | 80
Modified Full Analysis Set (mFAS) (All randomized subjects who received at least one dose of study treatment during the Treatment Period) | 77 | 76
Subjects Not Treated | 3 | 4
Main Study | 80 | 80
Mechanistic Sub-study | 36 | 0
Completed (Completed treatment) | 103 | 46
Not Completed | 13 | 34
Not completed — Adverse Event | 0 | 2
Not completed — Lack of Efficacy | 1 | 6
Not completed — Lost to Follow-up | 1 | 6
Not completed — Physician Decision | 0 | 1
Not completed — Subject/guardian decision | 8 | 15
Not completed — Subjects not treated | 3 | 4
Period: Follow-up Period
Arm/Group | Secukinumab 300 mg | Narrow-band Ultraviolet B (Nb-UVB)
Started | 73 (Subjects who entered follow-up period) | 39 (Subjects who entered follow-up period)
Main Study | 67 | 39
Mechanistic Sub-study | 6 | 0
Completed (Subjects in the Main Study who completed Week 104/208) | 13 | 8
Not Completed | 60 | 31
Not completed — Disease relapse | 32 | 7
Not completed — Lack of Efficacy | 1 | 2
Not completed — Lost to Follow-up | 4 | 6
Not completed — Physician Decision | 2 | 2
Not completed — Protocol Violation | 1 | 2
Not completed — Study terminated by Sponsor | 6 | 3
Not completed — Subject/guardian decision | 14 | 9

BASELINE CHARACTERISTICS:
Population: Subject disposition and baseline characteristics and presented using Randomized Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab 300 mg | Narrow-band Ultraviolet B (Nb-UVB) | Total
Number analyzed (Participants) | 116 | 80 | 196
Age, Customized [Count of Participants; unit: Participants]
  18 to 30 years | 56 | 30 | 86
  31 to 50 years | 60 | 50 | 110
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 25 | 60
  Male | 81 | 55 | 136
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1 | 1 | 2
  Asian | 2 | 3 | 5
  American Indian or Alaska Native | 0 | 1 | 1
  White | 113 | 72 | 185
  Unknown | 0 | 1 | 1
  Other | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Pain Assessment Severity Index (PASI) 90 at Week 52.
Description: The PASI quantifies the severity of a participant's psoriasis based on both "lesion severity" and the "percent of Body Surface Area (BSA)" affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI composite score varies in increments of 0.1 and range from 0 (no disease) to 72 (maximal disease), with higher scores representing greater severity of psoriasis. PASI 90 response is a binary measure defined as at least a 90% improvement in PASI score at Week 52, relative to baseline PASI score.
Time Frame: Baseline, Week 52
Population: Modified Full Analysis Set (mFAS) from the Main Study: all randomized subjects who received at least one dose of study treatment during the Treatment Period
Measure: Count of Participants; unit: Participants
Groups:
- Secukinumab 300 mg A1 (A1a+A1b): 80 patients (68 in Arm A1a and 12 in Arm A1b) with new-onset psoriasis will receive 300 mg secukinumab by subcutaneous (s.c.) injection at baseline, Weeks 1, 2, 3, 4 and then every 4 weeks until Week 48 inclusive (treatment duration = 52 weeks).
- Narrow-band Ultraviolet B (Nb-UVB) B1 (B1a+B1b): 80 patients (68 in Arm B1a and 12 in Arm B1b) with new-onset psoriasis received 1 or 2 cycles of narrow-band ultraviolet B (nb-UVB) of 12 weeks each with a maximum break of 28 weeks between cycles (patients with PASI 90 at Week 40 will not receive a second treatment cycle) (treatment duration = 52 weeks).
Arm/Group | Secukinumab 300 mg A1 (A1a+A1b) | Narrow-band Ultraviolet B (Nb-UVB) B1 (B1a+B1b)
Number analyzed (Participants) | 77 | 76
Participants | 70 | 32
Statistical Analysis 1: Comparison: Secukinumab 300 mg A1 (A1a+A1b) vs Narrow-band Ultraviolet B (Nb-UVB) B1 (B1a+B1b); Week 52 PASI 90; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 16.8, 95% CI 2-sided [5.9 to 48.3] — Logistic regression model with treatment as an explanatory variable and subset of significant covariates (including Baseline PASI score, age, BMI and their interaction terms with treatment) selected using forward selection method

2. Secondary Outcome: Number of Participants Who Achieved PASI 90 at Week 104
Description: The PASI quantifies the severity of a participant's psoriasis based on both "lesion severity" and the "percent of Body Surface Area (BSA)" affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI composite score varies in increments of 0.1 and range from 0 (no disease) to 72 (maximal disease), with higher scores representing greater severity of psoriasis. PASI 90 response is a binary measure defined as at least a 90% improvement in PASI score at Week 104, relative to baseline PASI score.
Time Frame: Baseline, Week 104
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 300 mg A1 (A1a+A1b) | Narrow-band Ultraviolet B (Nb-UVB) B1 (B1a+B1b)
Number analyzed (Participants) | 77 | 76
Participants | 23 | 26
Statistical Analysis 1: Comparison: Secukinumab 300 mg A1 (A1a+A1b) vs Narrow-band Ultraviolet B (Nb-UVB) B1 (B1a+B1b); Week 104 PASI 90; Test type: Superiority; p = 0.6530, Regression, Logistic; Odds Ratio (OR) = 0.8, 95% CI 2-sided [0.3 to 2.1] — Exact logistic regression method for Treatment group comparison, without using any covariates

3. Secondary Outcome: Number of Participants With IGA Mod 2011 0/1 Response at Week 52
Description: Investigators assessed the disease using the validated Investigator Global Assessment (IGA) mod 2011 and rated the disease from a score of 0 (clear skin) to 4 (severe disease). Response is defined as a score of 0 or 1 at Week 52.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Secukinumab 300 mg A1 (A1a+A1b) | Narrow-band Ultraviolet B (Nb-UVB) B1 (B1a+B1b)
Number analyzed (Participants) | 77 | 76
Percentage of participants | 85.7 [75.5 to 92.3] | 36.8 [26.3 to 48.7]

ADVERSE EVENTS:
Time Frame: On-treatment adverse events were collected from first dose of study treatment to 84 days after last dose of study medication (on-treatment), up to approximately 104 weeks. Evaluation of AEs and SAEs were repeated after dosing with study treatment (starting 85 days after last dose of treatment) until study termination notification.
Description: Any sign or symptom that occurred during the conduct of the trial and safety follow-up. The safety analysis were done for the Main Study and Mechanistic Sub-study in the safety population, which included all randomized subjects who received at least one dose of study medication. Patients were analyzed according to the actual treatment received.
Groups:
- Secukinumab 300 mg - On Treatment; Narrow-band Ultraviolet B (Nb-UVB) - On Treatment: AEs during on-treatment period (up to 84 days post-treatment)
- Secukinumab 300 mg - Post Treatment Follow-up; Narrow-band Ultraviolet B (Nb-UVB) - Post Treatment Follow-up: AEs during follow-up period (starting from 85 days post-treatment)
Arm/Group | Secukinumab 300 mg - On Treatment | Narrow-band Ultraviolet B (Nb-UVB) - On Treatment | Secukinumab 300 mg - Post Treatment Follow-up | Narrow-band Ultraviolet B (Nb-UVB) - Post Treatment Follow-up
All-Cause Mortality (participants affected / at risk) | 0/112 | 0/76 | 0/88 | 0/76
Serious Adverse Events (participants affected / at risk) | 6/112 | 1/76 | 0/88 | 1/76
Other Adverse Events (participants affected / at risk) | 29/112 | 8/76 | 7/88 | 2/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 300 mg - On Treatment (N=112) | Narrow-band Ultraviolet B (Nb-UVB) - On Treatment (N=76) | Secukinumab 300 mg - Post Treatment Follow-up (N=88) | Narrow-band Ultraviolet B (Nb-UVB) - Post Treatment Follow-up (N=76)
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Acute stress disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 300 mg - On Treatment (N=112) | Narrow-band Ultraviolet B (Nb-UVB) - On Treatment (N=76) | Secukinumab 300 mg - Post Treatment Follow-up (N=88) | Narrow-band Ultraviolet B (Nb-UVB) - Post Treatment Follow-up (N=76)
Nasopharyngitis (Infections and infestations) | 11 | 5 | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 8 | 2 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 0 | 5 | 1
Headache (Nervous system disorders) | 11 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/99/NCT03020199/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-18): https://cdn.clinicaltrials.gov/large-docs/99/NCT03020199/SAP_001.pdf